CLINICAL TRIAL: NCT04340648
Title: Measurement Algorithm Control and Optimization With Subsequent Performance Evaluation of the Vital USA GlucoseDetect™ During a Standardized Meal Test in Patients With Diabetes Mellitus Type 1 and Type 2
Brief Title: Measurement Algorithm Control, Optimization, and Performance Evaluation of the Vital USA GlucoseDetect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sciema UG (Other)
Responsible Party: Principal Investigator, Andreas Pfützner, Principle Investigator, Sciema UG
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VIT-NGM-001
Record Dates: First submitted 2020-03-23; First posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: patients are divided in two groups and both groups are enrolled sequential and undergo the same procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Vital GlucoseDetect — 11 time points for blood glucose measurements over 210 min including the ingestion of a standardized meal 30 min after the first blood glucose measurement.

SUMMARY:
Measurement Algorithm Control and Optimization with Subsequent Performance Evaluation of the Vital USA GlucoseDetect™ During a Standardized Meal Test in Patients with Diabetes mellitus Type 1 and Type 2

DETAILED DESCRIPTION:
This study is a combined, open label, prospective, comparative single-center study.

The study is separated in 3 consecutive study parts. The first 2 study parts include 16 patients each. In the third study part 16 additional patients will be enrolled. Study part 1 and 2 will be used for optimization and validation of the measurement algorithms of the Vital USA biosensor. During the third study part with enrolment of 16 additional patients, the precision and accuracy of the final Vital USA biosensor algorithm will be demonstrated. The visit schedule for all participants of all 3 study parts will be exactly the same. In all groups of participants, the Vital USA non-invasive monitoring biosensor will be individually introduced and assigned. During the experimental study visit, a standardized meal will be given to the participants. Before and after the standardized meal, glucose, heart rate, and pO2 will be measured using the Vital USA monitoring biosensor at time-points -30, 0, 15, 30, 45, 60, 75, 90, 120, 150 and 180 min. The glucose measurements will be compared to capillary blood glucose measurements by YSI Stat 2300. Parallel measurements of the heart rate and the pO2 using a patient monitor will be compared to the device readings.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 diabetic or healthy subject (50 % from each)
* Subjects who are able to complete informed consent form (by him/herself or by his/her guardian);
* 18 years old and above;
* Anatomically suitable finger in discretion of the investigator

Exclusion Criteria:

* Does not meet inclusion criteria;
* Any conditions that may hamper good visual contact between the finger or wrist and sensor, such as raised birthmarks, scars, tattoos;
* Pregnancy;
* Nursing mothers;
* Any skin scratch(es), damage, over dry, long nails on the measured finger;
* Unsuitable finger with the device might be excluded if recognized during the trial;
* Medication containing nitrates

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Performance and accuracy in glucose monitoring and other parameters | 210 min
  Performance and accuracy in monitoring glucose levels (in mg/dL) using the GlucoseDetect during a standardized meal experiment. Measurements (during the meal experiment) of the GlucoseDetectTM will be compared to the capillary blood glucose reference method YSI STAT 2300 (glucose in mg/dL).
Performance and accuracy in pO2 monitoring | 210 min
  Performance and accuracy in monitoring pO2 levels (in mmHg) using the GlucoseDetect during a standardized meal experiment. Measurements (during the meal experiment) of the GlucoseDetectTM will be compared to a patient monitor (pO2 (in mmHg).
Performance and accuracy in pulse monitoring | 210 min
  Performance and accuracy in monitoring the pulse (in beats/min) using the GlucoseDetect during a standardized meal experiment. Measurements (during the meal experiment) of the GlucoseDetectTM will be compared to a patient monitor (pulse (in beats/min).

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Pfützner, Prof. Dr. Dr., Principal Investigator — Pfützner Science & Health Institute GmbH
Locations (1):
- Pfützner Science & Health Institute GmbH, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No
the study will be summarized in a final report